CLINICAL TRIAL: NCT02067390
Title: Novel Urinary Biomarkers in the Detection of Vancomycin Associated Renal Injury
Brief Title: Urinary KIM-1 After Vancomycin or Linezolid Administration
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment
Sponsor: Midwestern University (Other)
Responsible Party: Principal Investigator, Marc Scheetz, Associate Professor, Midwestern University
Other Study IDs: STU00075251
Record Dates: First submitted 2014-02-13; First posted 2014-02-20 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vancomycin: Vancomycin
- Linezolid: Linezolid

SUMMARY:
Acute renal injury is a common complication of critical illness. Drug induced renal insult compounds the degree of injury in many patients, and a great deal of research has focused on prevention of this complication. Traditional biomarkers of renal injury like serum creatinine and blood urea nitrogen content fail to consistently predict harm among patients at risk. Kidney Injury Molecule 1 (KIM-1) will be studied as a biomarker of renal injury.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are male or female adults ≥18 years of age with an expected hospital stay of at least 48 hours.
* Eligible patients are already prescribed intravenous vancomycin or linezolid per their primary care providers as a standard of care and dosed in manner that is consistent with current institutional practices. Receipt of these antibiotics is not investigational.

Exclusion Criteria:

* Exclusion criteria will include patients who have stage 3or greater Chronic Kidney Disease or who have acute kidney injury prior to the start of intravenous vancomycin therapy, patients that only receive one dose of IV vancomycin or linezolid in total, as well as patients with potentially altered pharmacokinetic parameters (pregnant patients, burn patients, and those that are morbidly obese (BMI ≥ 40 kg/m2).
* Additionally, patients will be excluded if they are to receive more than 1 concurrent nephrotoxic medication within the prior 72 hours, have received intravenous contrast within 120 hours before randomization, exhibit baseline hematuria, or baseline proteinuria.
* A list of concurrent nephrotoxins that would exclude patients from the study is provided in Appendix C.
* Age Range: ≥18 years of age, if age > 90 will report as > 90 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically/Terminally Ill (ER, ICU)
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-09; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Urinary KIM-1 concentrations | Urinary levels from day -1 to day +5, clinical outcomes and variables followed for duration of hospitalization
  Urinary KIM-1 concentrations will be compared between patients receiving vancomycin and linezolid

CONTACTS AND LOCATIONS:
Overall Officials: Marc H Scheetz, PharmD, Principal Investigator — Northwestern Memorial Hospital / Midwestern University
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided